CLINICAL TRIAL: NCT01816139
Title: A Randomized, Multicenter, Double-Blind, Vehicle-Controlled Study to Evaluate the Safety and Efficacy of WC3011 in Postmenopausal Women
Brief Title: Multicenter Study to Evaluate Safety and Efficacy of WC3011 (Estradiol Vaginal Cream) in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR-05812
Record Dates: First submitted 2013-03-13; First posted 2013-03-21 (Estimated); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2021-09

CONDITIONS: Vulvovaginal Atrophy
Keywords: vaginal dryness; vaginal atrophy; estrogen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vehicle (2 Times/Week) (Experimental): Vehicle applied to the vagina daily for 2 weeks followed by dosing 2 times a week for 10 weeks.
  Interventions: Drug: Vehicle
- WC3011 Estradiol Vaginal Cream (2 Times/Week) (Placebo Comparator): WC3011 estradiol vaginal cream applied daily for 2 weeks followed by dosing 2 times a week for 10 weeks.
  Interventions: Drug: WC3011 Estradiol Vaginal Cream

INTERVENTIONS:
Drug: Vehicle — Vehicle Cream applied to the vagina daily for 2 weeks followed by dosing 2 times a week for 10 weeks
  Arms: Vehicle (2 Times/Week)
Drug: WC3011 Estradiol Vaginal Cream — WC3011 estradiol vaginal cream applied daily for 2 weeks followed by dosing 2 times a week for 10 weeks
  Arms: WC3011 Estradiol Vaginal Cream (2 Times/Week)

SUMMARY:
The primary objective of this study is to compare the efficacy of WC3011 with placebo vaginal gel in postmenopausal women for the relief of vaginal dryness caused by vaginal atrophy as measured by self-assessment, vaginal pH and vaginal smear.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Moderate to severe vaginal dryness
* Postmenopausal meeting one of the following: 12 months spontaneous amenorrhea, 6 months spontaneous amenorrhea with serum Follicle-stimulating hormone (FSH) > 40 milli-International Unit (mIU)/mL, 6 weeks postsurgical bilateral oophorectomy confirmed by surgical report, ultrasound or serum FSH > 40 mIU/mL, 6 weeks postsurgical hysterectomy with ovary failure confirmed by serum FSH > 40 mIU/mL
* Age ≥ 40 years or if bilateral oophorectomy ≥ 35 years
* Vaginal pH >5.0
* Less than or equal 5% superficial cells on vaginal wall cytologic smear
* Normal breast exam; if > 40 years, documentation of negative mammogram

Exclusion Criteria:

* Randomization in PR-04409, participation in clinical trial or use of investigational drug within 30 days prior to screening
* Smokes ≥ 15 cigarettes/day
* Known or suspected premalignant or malignant disease
* Cardiovascular disease, insulin-dependent diabetes mellitus, congestive heart failure, stroke or ischemic attack, thrombophlebitis or thromboembolic disorder
* Increased frequency/severity headaches with estrogen therapy
* Drug addiction/alcohol abuse within last 2 years
* Currently taking St. John's Wort or anticoagulant
* Uncontrolled hypertension or thyroid disorder, clinically significant depression or untreated urinary tract infection

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2013-11-19 (Actual); Study Completion 2013-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, PharmD, Study Director — Warner Chilcott
Locations (41):
- United States (41):
  - Warner Chilcott Investigational Study Site, Huntsville, Alabama
  - Warner Chilcott Investigational Study Site, Mobile, Alabama
  - Warner Chilcott Investigational Study Site, Phoenix, Arizona
  - Warner Chilcott Investigational Study Site, Scottsdale, Arizona
  - Warner Chilcott Investigational Study Site, Tucson, Arizona
  - Warner Chilcott Investigational Study Site, San Diego, California
  - Warner Chilcott Investigational Study Site, New London, Connecticut
  - Warner Chilcott Investigational Study Site, Boynton Beach, Florida
  - Warner Chilcott Investigational Study Site, Clearwater, Florida
  - Warner Chilcott Investigational Study Site, Jacksonville, Florida
  - Warner Chilcott Investigational Study Site, Miami, Florida
  - Warner Chilcott Investigational Study Site, Ormond Beach, Florida
  - Warner Chilcott Investigational Study Site, Palm Beach Gardens, Florida
  - Warner Chilcott Investigational Study Site, Pinellas Park, Florida
  - Warner Chilcott Investigational Study Site, West Palm Beach, Florida
  - Warner Chilcott Investigational Study Site, Atlanta, Georgia
  - Warner Chilcott Investigational Study Site, Roswell, Georgia
  - Warner Chilcott Investigational Study Site, Savannah, Georgia
  - Warner Chilcott Investigational Study Site, Granger, Indiana
  - Warner Chilcott Investigational Study Site, Marrero, Louisiana
  - Warner Chilcott Investigational Study Site, New Orleans, Louisiana
  - Warner Chilcott Investigational Study Site, Kalamazoo, Michigan
  - Warner Chilcott Investigational Study Site, Las Vegas, Nevada
  - Warner Chilcott Investigational Study Site, Moorestown, New Jersey
  - Warner Chilcott Investigational Study Site, Greensboro, North Carolina
  - Warner Chilcott Investigational Study Site, New Bern, North Carolina
  - Warner Chilcott Investigational Study Site, Winston-Salem, North Carolina
  - Warner Chilcott Investigational Study Site, Cleveland, Ohio
  - Warner Chilcott Investigational Study Site, Columbus, Ohio
  - Warner Chilcott Investigational Study Site, Jenkintown, Pennsylvania
  - Warner Chilcott Investigational Study Site, Philadelphia, Pennsylvania
  - Warner Chilcott Investigational Study Site, Pittsburgh, Pennsylvania
  - Warner Chilcott Investigational Study Site, Bluffton, South Carolina
  - Warner Chilcott Investigational Study Site, Dallas, Texas
  - Warner Chilcott Investigational Study Site, Houston, Texas
  - Warner Chilcott Investigational Study Site, San Antonio, Texas
  - Warner Chilcott Investigational Study Site, Salt Lake City, Utah
  - Warner Chilcott Investigational Study Site, Norfolk, Virginia
  - Warner Chilcott Investigational Study Site, Richmond, Virginia
  - Warner Chilcott Investigational Study Site, Seattle, Washington
  - Warner Chilcott Investigational Study Site, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (2 Times/Week)
Started | 289 | 287
Safety Population | 287 | 286
Modified Intent-to-treat (mITT) Population | 240 | 248
Completed | 261 | 265
Not Completed | 28 | 22
Not completed — Adverse Event | 6 | 8
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrew Consent | 6 | 4
Not completed — Protocol Violation | 6 | 3
Not completed — Reason not Specified | 4 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who were randomized into the study and took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (2 Times/Week) | Total
Number analyzed (Participants) | 287 | 286 | 573
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (6.1) | 59.5 (6.7) | 59.6 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 287 | 286 | 573
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Participant's Self-Assessment of Severity of Vaginal Dryness to Final Assessment
Description: Participant's self-assessment of Vaginal Dryness was scored on a 4-point scale where: 0=none, 1=mild, 2=moderate or 3=severe. Higher scores indicate the most bothersome symptoms. A negative change from Baseline indicates improvement. Final assessment is defined as the last available postbaseline assessment.
Time Frame: Baseline (Day 0) to final assessment (Up to Week 12)
Population: Modified Intent-to-Treat (mITT) Population included participants in safety population who had at least 1 postbaseline primary efficacy assessment and had: ≤5% superficial cells on a vaginal wall smear, a vaginal pH >5.0 and participant's most bothersome symptom of VVA was vaginal dryness with moderate to severe intensity. Number analyzed is the number of participants with available data at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (2 Times/Week)
Number analyzed (Participants) | 240 | 248
score on a scale
  Baseline | 2.5 (0.50) | 2.5 (0.50)
  Change from Baseline to Final Assessment: number analyzed (Participants) | 240 | 247
  Change from Baseline to Final Assessment | -1.2 (0.92) | -1.4 (0.94)

2. Primary Outcome: Change From Baseline in Vaginal pH to Final Assessment
Description: Vaginal pH was obtained at baseline and final visit of the study. The pH was a numeric value from 0 to 14 expressing the acidity or alkalinity of the vaginal fluids where 7 was neutral, lower values were more acidic (values of 0-6) and higher values more alkaline (values of 8-14). A negative change from Baseline indicates improvement. Final assessment is defined as the last available postbaseline assessment.
Time Frame: Baseline (Day 0) to final assessment (Up to Week 12)
Population: mITT Population included participants in safety population who had at least 1 postbaseline primary efficacy assessment and had: ≤5% superficial cells on a vaginal wall smear, a vaginal pH >5.0 and participant's most bothersome symptom of VVA was vaginal dryness with moderate to severe intensity. Number analyzed is the number of participants with available data at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (2 Times/Week)
Number analyzed (Participants) | 240 | 248
score on a scale
  Baseline | 6.33 (0.65) | 6.34 (0.65)
  Change from Baseline to Final Assessment: number analyzed (Participants) | 231 | 244
  Change from Baseline to Final Assessment | -0.31 (0.80) | -1.26 (0.99)

3. Primary Outcome: Change From Baseline in the Percentage of Vaginal Superficial Cells to Final Assessment
Description: Vaginal wall smears were collected from each participant. The smears were sent to the central laboratory for analysis to determine the percentage of superficial cells. A positive change from Baseline indicates improvement. Final assessment is defined as the last available postbaseline assessment.
Time Frame: Baseline (Day 0) to final assessment (Up to Week 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (2 Times/Week)
Number analyzed (Participants) | 240 | 248
percentage of superficial cells
  Baseline | 0.3 (1.05) | 0.4 (1.13)
  Change from Baseline to Final Assessment: number analyzed (Participants) | 228 | 235
  Change from Baseline to Final Assessment | 0.8 (5.68) | 8.6 (14.49)

4. Primary Outcome: Change From Baseline in the Percentage of Vaginal Parabasal Cells to Final Assessment
Description: Vaginal wall smears were collected from each participant. The smears were sent to the central laboratory for analysis to determine the percentage of parabasal cells. A negative change from Baseline indicates improvement. Final assessment is defined as the last available postbaseline assessment.
Time Frame: Baseline (Day 0) to final assessment (Up to Week 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (2 Times/Week)
Number analyzed (Participants) | 240 | 248
percentage of parabasal cells
  Baseline | 46.5 (44.81) | 44.2 (42.29)
  Change from Baseline to Final Assessment: number analyzed (Participants) | 228 | 235
  Change from Baseline to Final Assessment | -4.4 (42.93) | -37.4 (42.62)

5. Secondary Outcome: Change From Baseline in Participant's Self-Assessment of Severity of Vaginal Dryness to Weeks 2, 4, 8, and 12
Description: Participant's self-assessment of Vaginal Dryness was scored on a 4-point scale where: 0=none, 1=mild, 2=moderate or 3=severe. Higher scores indicate the most bothersome symptoms. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Weeks 2, 4, 8, and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (2 Times/Week)
Number analyzed (Participants) | 240 | 248
score on a scale
  Baseline | 2.5 (0.50) | 2.5 (0.50)
  Change from Baseline to Week 2: number analyzed (Participants) | 236 | 247
  Change from Baseline to Week 2 | -0.9 (0.92) | -1.0 (0.94)
  Change from Baseline to Week 4: number analyzed (Participants) | 229 | 239
  Change from Baseline to Week 4 | -1.1 (0.87) | -1.2 (0.86)
  Change from Baseline to Week 8: number analyzed (Participants) | 228 | 233
  Change from Baseline to Week 8 | -1.2 (0.87) | -1.4 (0.85)
  Change from Baseline to Week 12: number analyzed (Participants) | 224 | 232
  Change from Baseline to Week 12 | -1.2 (0.90) | -1.5 (0.93)

6. Secondary Outcome: Change From Baseline in Participants Self-Assessment of the Symptoms of VVA
Description: Self-Assessment of the symptoms of VVA (vaginal and/or vulvar irritation/ Itching, dysuria, and dyspareunia) were evaluated by a questionnaire. Each symptom was scored on a 4-point scale where: 0=none, 1=mild, 2=moderate, or 3=severe. Higher scores indicate the most bothersome symptoms. A negative change from Baseline indicates improvement. Final Assessment is defined as the last available post-baseline assessment for the given efficacy endpoint.
Time Frame: Baseline (Day 0) to Weeks 2, 4, 8, 12 and Final Assessment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (2 Times/Week)
Number analyzed (Participants) | 240 | 248
score on a scale
  Vaginal Itching - Baseline | 1.1 (0.97) | 1.1 (0.97)
  Vaginal Itching - Change from Baseline to Week 2: number analyzed (Participants) | 235 | 247
  Vaginal Itching - Change from Baseline to Week 2 | -0.5 (0.93) | -0.5 (0.95)
  Vaginal Itching - Change from Baseline to Week 4: number analyzed (Participants) | 229 | 239
  Vaginal Itching - Change from Baseline to Week 4 | -0.6 (0.99) | -0.6 (0.89)
  Vaginal Itching - Change from Baseline to Week 8: number analyzed (Participants) | 228 | 233
  Vaginal Itching - Change from Baseline to Week 8 | -0.6 (0.95) | -0.6 (0.92)
  Vaginal Itching - Change from Baseline to Week 12: number analyzed (Participants) | 224 | 232
  Vaginal Itching - Change from Baseline to Week 12 | -0.7 (1.00) | -0.7 (0.94)
  Vaginal Itching - Change from Baseline to Final Assessment: number analyzed (Participants) | 240 | 247
  Vaginal Itching - Change from Baseline to Final Assessment | -0.7 (0.99) | -0.6 (0.99)
  Dysuria - Baseline | 0.3 (0.66) | 0.4 (0.72)
  Dysuria - Change from Baseline to Week 2: number analyzed (Participants) | 236 | 247
  Dysuria - Change from Baseline to Week 2 | -0.1 (0.71) | -0.2 (0.66)
  Dysuria - Change from Baseline to Week 4: number analyzed (Participants) | 229 | 239
  Dysuria - Change from Baseline to Week 4 | -0.1 (0.75) | -0.2 (0.69)
  Dysuria - Change from Baseline to Week 8: number analyzed (Participants) | 228 | 233
  Dysuria - Change from Baseline to Week 8 | -0.2 (0.65) | -0.2 (0.75)
  Dysuria - Change from Baseline to Week 12: number analyzed (Participants) | 224 | 232
  Dysuria - Change from Baseline to Week 12 | -0.2 (0.65) | -0.2 (0.69)
  Dysuria - Change from Baseline to Final Assessment: number analyzed (Participants) | 240 | 247
  Dysuria - Change from Baseline to Final Assessment | -0.2 (0.64) | -0.2 (0.71)
  Dyspareunia - Baseline: number analyzed (Participants) | 186 | 181
  Dyspareunia - Baseline | 2.1 (0.92) | 2.1 (0.99)
  Dyspareunia - Change from Baseline to Week 2: number analyzed (Participants) | 128 | 129
  Dyspareunia - Change from Baseline to Week 2 | -0.7 (0.91) | -0.7 (1.04)
  Dyspareunia - Change from Baseline to Week 4: number analyzed (Participants) | 128 | 129
  Dyspareunia - Change from Baseline to Week 4 | -1.0 (0.90) | -1.1 (1.05)
  Dyspareunia - Change from Baseline to Week 8: number analyzed (Participants) | 133 | 127
  Dyspareunia - Change from Baseline to Week 8 | -0.9 (0.99) | -1.2 (1.03)
  Dyspareunia - Change from Baseline to Week 12: number analyzed (Participants) | 134 | 130
  Dyspareunia - Change from Baseline to Week 12 | -1.1 (0.97) | -1.1 (1.12)
  Dyspareunia - Change from Baseline to Final Assessment: number analyzed (Participants) | 154 | 151
  Dyspareunia - Change from Baseline to Final Assessment | -1.0 (0.95) | -1.1 (1.11)

7. Secondary Outcome: Percentage of Participants With Vaginal Bleeding Associated With Sexual Activity
Description: Vaginal bleeding associated with sexual activity was assessed by participants as either "present" or "absent". Number of participants with assessment "present" are reported. Final assessment is defined as the last available postbaseline assessment.
Time Frame: Baseline (Day 0) and Weeks 2, 4, 8, 12 and Final Assessment
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (2 Times/Week)
Number analyzed (Participants) | 184 | 177
percentage of participants
  Baseline | 18.5 | 24.3
  Week 2: number analyzed (Participants) | 131 | 131
  Week 2 | 8.4 | 8.4
  Week 4: number analyzed (Participants) | 131 | 130
  Week 4 | 6.1 | 4.6
  Week 8: number analyzed (Participants) | 137 | 134
  Week 8 | 8.0 | 6.7
  Week 12: number analyzed (Participants) | 137 | 133
  Week 12 | 6.6 | 3.8
  Final Assessment: number analyzed (Participants) | 164 | 158
  Final Assessment | 7.9 | 5.1

8. Secondary Outcome: Change From Baseline in the Investigator's Assessment of Each of the Signs of VVA to Week 12 and Final Assessment
Description: Investigator's assessment of vaginal health was performed by visual inspection of the vagina with respect to the signs of VVA: atrophy, pallor, vaginal dryness, friability, and petechiae each graded on a 4-point scale where: 0=none, 1=mild, 2=moderate or 3=severe. Higher scores are worse. A negative change from Baseline indicates improvement. Final assessment is defined as the last available postbaseline assessment.
Time Frame: Baseline (Day 0) to Week 12 and Final Assessment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (2 Times/Week)
Number analyzed (Participants) | 240 | 248
score on a scale
  Atrophy - Baseline | 2.1 (0.60) | 2.0 (0.65)
  Atrophy - Change from Baseline to Week 12: number analyzed (Participants) | 224 | 231
  Atrophy - Change from Baseline to Week 12 | -0.4 (0.74) | -0.7 (0.80)
  Atrophy - Change from Baseline to Final Assessment: number analyzed (Participants) | 231 | 244
  Atrophy - Change from Baseline to Final Assessment | -0.4 (0.74) | -0.7 (0.79)
  Pallor - Baseline | 1.9 (0.67) | 1.9 (0.66)
  Pallor - Change from Baseline to Week 12: number analyzed (Participants) | 224 | 231
  Pallor - Change from Baseline to Week 12 | -0.4 (0.79) | -0.9 (0.79)
  Pallor - Change from Baseline to Final Assessment: number analyzed (Participants) | 231 | 244
  Pallor - Change from Baseline to Final Assessment | -0.4 (0.79) | -0.9 (0.82)
  Dryness - Baseline | 2.0 (0.65) | 2.0 (0.69)
  Dryness - Change from Baseline to Week 12: number analyzed (Participants) | 224 | 231
  Dryness - Change from Baseline to Week 12 | -0.6 (0.84) | -1.1 (0.89)
  Dryness - Change from Baseline to Final Assessment: number analyzed (Participants) | 231 | 244
  Dryness - Change from Baseline to Final Assessment | -0.6 (0.84) | -1.1 (0.89)
  Friability - Baseline | 1.1 (0.86) | 1.1 (0.86)
  Friability - Change from Baseline to Week 12: number analyzed (Participants) | 224 | 231
  Friability - Change from Baseline to Week 12 | -0.5 (0.81) | -0.8 (0.92)
  Friability - Change from Baseline to Final Assessment: number analyzed (Participants) | 231 | 244
  Friability - Change from Baseline to Final Assessment | -0.5 (0.81) | -0.8 (0.92)
  Petechiae - Baseline | 0.8 (0.86) | 0.8 (0.82)
  Petechiae - Change from Baseline to Week 12: number analyzed (Participants) | 224 | 231
  Petechiae - Change from Baseline to Week 12 | -0.4 (0.71) | -0.6 (0.82)
  Petechiae - Change from Baseline to Final Assessment: number analyzed (Participants) | 231 | 244
  Petechiae - Change from Baseline to Final Assessment | -0.4 (0.74) | -0.6 (0.83)

9. Secondary Outcome: Change From Baseline in the Percentage of Vaginal Superficial Cells to Week 12
Description: Vaginal wall smears were collected from each participant. The smears were sent to the central laboratory for analysis to determine the percentage of superficial cells. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (2 Times/Week)
Number analyzed (Participants) | 240 | 248
percentage of superficial cells
  Baseline | 0.3 (1.05) | 0.4 (1.13)
  Change from Baseline to Week 12: number analyzed (Participants) | 222 | 216
  Change from Baseline to Week 12 | 0.6 (3.35) | 9.3 (14.87)

10. Secondary Outcome: Change From Baseline in the Percentage of Vaginal Parabasal Cells to Week 12
Description: Vaginal wall smears were collected from each participant. The smears were sent to the central laboratory for analysis to determine the percentage of parabasal cells. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (2 Times/Week)
Number analyzed (Participants) | 240 | 248
percentage of parabasal cells
  Baseline | 46.5 (44.81) | 44.2 (42.29)
  Change from Baseline to Week 12: number analyzed (Participants) | 222 | 216
  Change from Baseline to Week 12 | -4.7 (43.39) | -38.7 (41.58)

ADVERSE EVENTS:
Time Frame: From first dose through the last study visit (Up to 12 weeks)
Description: Safety Population included all participants who were randomized into the study and took at least 1 dose of study drug.
Arm/Group | Vehicle (2 Times/Week) | WC3011 Estradiol Vaginal Cream (2 Times/Week)
All-Cause Mortality (participants affected / at risk) | 0/287 | 0/286
Serious Adverse Events (participants affected / at risk) | 2/287 | 2/286
Other Adverse Events (participants affected / at risk) | 35/287 | 38/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (2 Times/Week) (N=287) | WC3011 Estradiol Vaginal Cream (2 Times/Week) (N=286)
Myocardial Infarction (Cardiac disorders) | 0 | 1
Hiatus Hernia (Gastrointestinal disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Postoperative Wound Infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (2 Times/Week) (N=287) | WC3011 Estradiol Vaginal Cream (2 Times/Week) (N=286)
Urinary tract infection (Infections and infestations) | 17 | 15
Application site pain (General disorders) | 16 | 9
Vulvovaginal mycotic infection (Infections and infestations) | 3 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.